CLINICAL TRIAL: NCT05019352
Title: Cytokine Adsorption in Patients With Acute-on-chronic Liver Failure (CYTOHEP) - a Single Center, Open-label, Randomized, Controlled Intervention Trial
Brief Title: Cytokine Adsorption in Acute-on-chronic Liver Failure
Acronym: CYTOHEP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dr. Alexander Supady (Other)
Responsible Party: Sponsor-Investigator, Dr. Alexander Supady, Oberarzt - Attending Physician, University Hospital Freiburg
Organization: University Hospital Freiburg (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CYTOHEP
Record Dates: First submitted 2021-08-17; First posted 2021-08-24 (Actual); Last update posted 2021-11-02 (Actual); Status verified 2021-10

CONDITIONS: Acute-On-Chronic Liver Failure; Renal Failure
Keywords: cytokine adsorption; renal replacement therapy; interleukins; cytokines
MeSH Terms: conditions — Acute-On-Chronic Liver Failure; Renal Insufficiency

STUDY DESIGN:
Intervention Model Description: In a prallel design participants will be randomly assigned to three different trial groups
Masking Description: open-label trial without masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CRRT with cytokine adsorption (Experimental): Patients will be treated with CRRT and extracorporeal hemoadsorption for 72 hours
  Interventions: Device: CytoSorb cytokine adsorber; Device: CRRT
- CRRT without cytokine adsorption (Experimental): Patients will be treated with CRRT without extracorporeal hemoadsorption for 72 hours
  Interventions: Device: CRRT
- no CRRT, no cytokine adsorption (No Intervention): Patients will not receive CRRT, nor extracorporeal hemoadsorption. CRRT will only be initiated in case of severe electrolyte disorders or unmanageable fluid overload

INTERVENTIONS:
Device: CytoSorb cytokine adsorber — device for extracorporeal hemoadsorption
  Arms: CRRT with cytokine adsorption
Device: CRRT — continuous renal replacement therapy
  Arms: CRRT with cytokine adsorption; CRRT without cytokine adsorption

SUMMARY:
The CYTOHEP study is a prospective, randomized, single center, open-label, controlled intervention trial to assess the benefit of extracorporeal hemoadsorption using the CytoSorb device in patients with acute-on-chronic liver failure. The primary goal for this trial is to assess whether the CytoSorb device used in addition to continuous renal replacement therapy (CRRT) will be able to significantly reduce bilirubin in the patient blood as compared to the control group treated with CRRT alone (i.e., without extracorporeal hemoadsorption).

The rationale for this study is based on considerations about the role of systemic inflammation in acute decompensation of liver cirrhosis and ACLF, in-vitro data of the effectiveness CytoSorb for the removal of molecules with a pathophysiological role in acute-on-chronic liver failure, and recent reports on the successful use of extracorporeal hemoadsorption in combination with CRRT in critically ill patients with acute liver dysfunction.

DETAILED DESCRIPTION:
Liver cirrhosis is a major healthcare problem. The clinical course of cirrhosis can be separated in compensated and decompensated cirrhosis. Patients with compensated cirrhosis are largely asymptomatic and the development of decompensating events is a major hallmark in the course of the disease as median survival decreases from 12 years to less than 2 years. The development of extrahepatic organ complications in decompensated cirrhosis has been identified as a major prognostic milestone and has been described as acute-on-chronic liver failure (ACLF). ACLF is understood as a dynamic process and may evolve within days leading to multi-organ failure with renal failure being the most common organ involvement (56%), followed by liver and coagulation failure (44% and 28%, respectively). ACLF is associated with a high 28-day mortality.

During recent years, systemic inflammation has been recognized as a major driver of hepatic decompensation and progression of liver cirrhosis to ACLF. Importantly, systemic inflammation was described as an important trigger for development of extrahepatic organ failures, such as renal failure, development of hepatopulmonary syndrome, cirrhotic cardiomyopathy and hepatic encephalopathy. Systemic inflammation is particularly relevant in the pathogenesis of acute hepatic decompensation and is also associated with reduced survival. Therefore, elimination of drivers of inflammatory response and inflammatory cytokines in addition to established therapeutic approaches aiming at a reduction of bacterial translocation and mitigation of portal hypertension may help control excessive inflammatory activity and thus support hepatic recompensation. Previous in-vitro examinations and studies in non-cirrhotic inflammatory disorders have shown that proinflammatory cytokines and other factors can effectively be removed by extracorporeal hemoadsorption in the CytoSorb adsorber.

The CYTOHEP study is designed as a prospective, randomized, single center, open-label, controlled intervention trial to assess the benefit of extracorporeal hemoadsorption using the CytoSorb device in patients with acute-on-chronic liver failure. The primary goal for this pilot trial is to assess whether the CytoSorb device used in addition to CRRT will be able to significantly reduce bilirubin in the patient blood as compared to the control group treated with CRRT alone (i.e., without extracorporeal hemoadsorption).

Within this trial, CRRT will be initiated early, i.e., in patients with acute kidney injury (AKI) Kidney Disease: Improving Global Outcome (KDIGO) stage 3. For safety assessment, a third group will be assessed without early initiation of CRRT and extracorporeal hemoadsorption. After trial inclusion, all patients will be randomized in a 1:1:1 fashion in one of the study groups.

ELIGIBILITY:
Inclusion Criteria:

* adult patients (≥ 18 years) admitted to the University Medical Center Freiburg, Germany
* acute-on-chronic liver failure (ACLF) WITH acute kidney injury according to Kidney Disease: Improving Global Outcome (KDIGO) criteria stage 3 (≥ 3-fold increase of serum creatinine OR increase of serum creatinine to ≥ 4 mg/dl OR urine output ≤ 0.3 ml/kg/h for ≥ 24 hours OR anuria for ≥ 12 hours) AND serum bilirubin ≥ 5 mg/dl

Exclusion Criteria:

* known patient will against participation in the study or against the measures applied in the study
* a decision made prior to inclusion to stop further treatment of the patient within the next 24 hours
* no complete remission of malignancy including hepatocellular carcinoma within the past 12 months
* patients on the waiting list for liver transplant or the potential option for being listed for liver transplant within the next 6 months
* liver cirrhosis in patients after liver transplantation
* ongoing intermittent or continuous renal replacement therapy before study inclusion

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Estimated)
Dates: Start 2021-10-25 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-01-30 (Estimated)

PRIMARY OUTCOMES:
Serum bilirubin | 72 hours
  Serum bilirubin after 72 hours

SECONDARY OUTCOMES:
Survival time | 30 days
  Survival time from baseline
Interleukin-6 | 72 hours
  Interleukin-6 after 72 hours
Liver function parameters | 72 hours
  Quick/INR, AST, ALT, AP, g-GT
Blood lactate | 72 hours
  Lactate concentration after 72 hours
CLIF-SOFA-score | 72 hours
  CLIF-SOFA-score
MELD score | 72 hours
  MELD score
SOFA score | 72 hours
  SOFA score
SAPS II | 72 hours
  SAPS II
FIPS score | 72 hours
  FIPS score
Ventilator free days | 30 days
  Ventilator free days (VeFD) in the first 30 days after randomization, where each day on invasive mechanical ventilation (IMV), non-invasive ventilation (NIV), or ECMO is defined as ventilator day. VeFD=0, if the patient dies in the first 30 days after randomization
vasopressor dosage | 72 hours
  dosage of epinephrine, norepinephrine, dobutamine, argipressin and terlipressin
Vasopressor free days | 30 days
  Vasopressor free days (VaFD) in the first 30 days after randomization, where each day with any dose of epinephrine, norepinephrine, dobutamine, argipressin or terlipressin is defined as vasopressor day. VaFD=0, if the patient dies in the first 30 days after randomization
Dialysis free days | 30 days
  Dialysis free days (DFD) in the first 30 days after randomization, where each day on renal replacement therapy (RRT) is defined as dialysis day. DFD=0, if the patient dies in the first 30 days after randomization
Inflammatory biomarkers | 72 hours
  A biomarker panel of pro- and anti-inflammatory cytokines (blood samples will be frozen and stored for later analyses, panel will be determined at the time of analysis)

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Supady, MD, MPH, Principal Investigator — University Hospital Freiburg
Locations (1):
- University Clinic Freiburg, Freiburg im Breisgau, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sekandarzad A, Weber E, Prager EP, Graf E, Bettinger D, Wengenmayer T, Supady A. Cytokine adsorption in patients with acute-on-chronic liver failure (CYTOHEP)-a single center, open-label, three-arm, randomized, controlled intervention trial. Trials. 2022 Mar 18;23(1):222. doi: 10.1186/s13063-022-06139-6. PMID 35303938